CLINICAL TRIAL: NCT03485937
Title: Impact of Pre-Operative Videos on Mohs Surgery Patient Anxiety and Satisfaction
Brief Title: Impact of Videos on Patient Anxiety and Satisfaction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: low accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE1618
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Mohs Surgery
Keywords: anxiety; patient satisfaction; video education; skin cancer; linear closure on the face
MeSH Terms: conditions — Anxiety Disorders; Patient Satisfaction; Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Operative Videos + verbal/written instructions (Experimental): This video contains the same instructions that the patient receives when they arrive at the clinic, as well as a video walk through of the clinic/patient room. Videos will be created by the study team to ensure that the content coincides with what is delivered in the standard-of-care verbal and written instructions.
  Interventions: Behavioral: Pre-Operative Videos; Behavioral: verbal instructions; Behavioral: written instructions
- verbal/written instructions (Active Comparator): This arm will receive the standard-of-care verbal/written instructions and the pre-operative video explanation. These instructions contain the same content as in the pre-operative videos
  Interventions: Behavioral: verbal instructions; Behavioral: written instructions

INTERVENTIONS:
Behavioral: Pre-Operative Videos — Videos will be created by the study team to ensure that the content coincides with what is delivered in the standard-of-care verbal and written instructions. The videos will be split into two modules: 1) preparing for Mohs Surgery 2) Mohs Surgery Walk through. The intervention, in the form of a video walk through, will be provided to the patient via email prior to their surgical procedure once they schedule an appointment with the Mohs clinic for their surgery day.
  Arms: Pre-Operative Videos + verbal/written instructions
Behavioral: verbal instructions — As part of the standard of care for patients receiving Mohs surgery, patients are told about the day of their surgery and what to expect
Behavioral: written instructions — As part of the standard of care for patients receiving Mohs surgery, patients receive written material about the day of their surgery and what to expect

SUMMARY:
The purpose of this research is to look at how educational videos might affect patient satisfaction and anxiety before Mohs surgery day. Patients will be randomized to either: 1) a group that receives educational videos before the visit in addition to standard-of-care written and verbal instructions OR 2) a group that receives only standard-of-care written and verbal instructions.

DETAILED DESCRIPTION:
The primary objective of this study is to determine if pre-operative videos describing the patient's forthcoming day in the Mohs clinic decrease pre-operative patient anxiety and increase postoperative patient satisfaction, when added to standard of care written and verbal instruction.

Design/Study Type This study will be a randomized control trial in which patients will be randomized to either the intervention (pre-operative Mohs Surgery video viewing) or control (standard of care) group in order to understand the impact of the video on patient anxiety and satisfaction. Patients will be randomized using an Accelerated Biased Coin Design in the statistical program R.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at the University Hospitals Cleveland Medical Center Mohs Clinic to undergo a linear closure on the face.
* Fluent English speakers

Exclusion Criteria:

* Non-fluent English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Difference in mean Likert scale rating of subject satisfaction score | Up to 8 weeks after visit
  For subject satisfaction score, the mean Likert scale rating for the control and intervention groups will be compared. The scale being used is a six item instrument with individual scores ranging from 1-5 (total score 6-30). Higher scores indicate greater satisfaction.
Difference in mean Likert scale rating of subject anxiety score | Up to 8 weeks after visit
  For subject anxiety score, the mean Likert scale rating for the control and intervention groups will be compared. The scale being used is a seven item instrument with individual scores ranging from 1-5 with positive worded items scored in reverse (total score 7-35). Higher scores indicate greater anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy S. Bordeaux, MD, MPH, Principal Investigator — University Hospitals, Case Comprehensive Cancer Center